CLINICAL TRIAL: NCT05279209
Title: Catheter-directed Sclerotherapy Versus Surgical Resecction: Randomized Controlled Trial Comparing Ovarian Function and Therapeutic Efficacy After Treatment of Ovarian Endometrioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2021-1512
Record Dates: First submitted 2022-01-11; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Endometrioma
Keywords: Endometrioma; resection; enucleation; sclerotherapy; ovarian function
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sclerotherapy (Experimental): Patients who receive uterine artery embolization for symptomatic fibroids
  Interventions: Procedure: catheter-directed sclerotherapy
- Surgery (Active Comparator): Patients who receive uterine artery embolization for symptomatic fibroids
  Interventions: Procedure: surgical resection

INTERVENTIONS:
Procedure: catheter-directed sclerotherapy — Ovarian endometrioma is targeted under transvaginal/transabdominal ultrasound. A guidewire is inserted to the lesion and is exchanged for a catheter. The cystic content is thoroughly aspirated and then sclerotherapy is performed by injecting 99% ethanol.
  Arms: Sclerotherapy
Procedure: surgical resection — Surgical resection of the ovarian endometrioma is performed under general anesthesia. To preserve the residual ovarian function, enucleation is the primary surgical technique.
  Arms: Surgery

SUMMARY:
The primary purpose of this study is to compare residual ovarian function and therapeutic efficacy of surgical resection and catheter-directed sclerotherapy for ovarian endometrioma

DETAILED DESCRIPTION:
Screening

* History, Physical examination
* Vital signs
* Laboratory test (Serum AMH, CA-125, HE-4) / EKG / MRI
* EHP-30

Intervention

* Surgical enucleation or catheter-directed sclerotherapy
* Laboratory test / EKG
* Adverse event monitoring

Follow-up visit #1 (1 month)

* Vital signs
* Lab test (AMH, CA-125) / Ultrasound
* Adverse event monitoring

Follow-up visit #2 (6 months)

* Vital signs
* Lab test (AMH, CA-125) / Ultrasound / Contrast-enhanced MRI
* EHP-30

Follow-up visit #3 (12months)

* Vital signs
* Lab test (AMH, CA-125) / Ultrasound
* EHP-30

ELIGIBILITY:
Inclusion Criteria:

1. Women with symptomatic fibroids (age: 20 - 60 years old)

Exclusion Criteria:

1. Gynecologic malignancy
2. Ongoing infection or inflammation
3. Coagulopathy (platelet < 50,000 or INR > 1.5)
4. Extraovarian endometriosis
5. Serum AMH of 5 or higher
6. Drug allergy
7. Illiteracy
8. Pregnancy

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-12-18 (Actual); Primary Completion 2022-12-17 (Estimated); Study Completion 2023-12-17 (Estimated)

PRIMARY OUTCOMES:
Serum AMH | Serum AMH at 1month after catheter-directed sclerotherapy
  Serum AMH: A measure of ovarian function
Serum AMH | Serum AMH at 6months after catheter-directed sclerotherapy
  Serum AMH: A measure of ovarian function
Serum AMH | Serum AMH at 12 months after catheter-directed sclerotherapy
  Serum AMH: A measure of ovarian function

SECONDARY OUTCOMES:
Recurrence | 1, 6, and 12 months
  Recurrence of symptoms or development of ovarian endometrioma of 2cm or larger on follow-up imaging (surgery) vs. Recurrence of symptoms or detection of the lesion 50% or larger to the size of the initial lesion on follow-up imaging (sclerotherapy).
hospital stay | duration of admission (days), up to 5 days
  Time from admission to discharge
serum CA-125 | 1, 6, 12 months
  Serum CA-125 (unit/mL): Surrogate marker for therapeutic efficacy (A reduction in serum CA-125 represents a response to the intervention)
EHP-30 (Endometriosis Health Profile-30) | 6 and 12 months
  EHP-30: A measure of quality of life related to ovarian endometrioma (Scale of 0 to 30, A higher score represents adverse impact of daily living by the endometriosis)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No